CLINICAL TRIAL: NCT05685004
Title: Randomized Phase 2b Study of Safety And Efficacy Of TVI-Brain-1 Combined With Conformal Radiotherapy And Temozolomide Vs Standard Therapy In Newly Diagnosed MGMT Negative Glioblastoma Multiforme (GBM)
Brief Title: Study of Neoantigen-specific Adoptive T Cell Therapy for Newly Diagnosed MGMT Negative Glioblastoma Multiforme (GBM)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TVAX Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TVI-AST-008
Record Dates: First submitted 2022-12-22; First posted 2023-01-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma Multiforme of Brain
MeSH Terms: interventions — Standard of Care; Radiotherapy; Temozolomide; Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded over-read of sequential MRI assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Subjects will have standard surgery which will be followed approximately 5 weeks later by combined radiotherapy and chemotherapy consisting of temozolomide 75 mg/m2 dosed once daily beginning on the first day of radiotherapy and continuing until the final day of radiotherapy. Subjects will receive adjuvant temozolomide, and proceed with post therapy surveillance.
  Interventions: Procedure: Standard of Care; Radiation: Radiotherapy; Drug: Temozolomide
- Interventional TVI-Brain-1 Autologous Vaccine and activated autologous blood-derived t cells (Experimental): TVI-Brain-1 immunotherapy is integrated with radiation and temozolomide in the test group in the following manner: 1) Subjects undergo surgical resection of their cancer and are tapered off steroids. 2) Subjects receive the first vaccination of TVI-Brain-1 as soon as the laboratory prepared vaccine is available for use (approximately 7 - 14 days following surgery). 3) Subjects receive a second vaccination 7-10 days later. 4) Subjects are leukapheresed to obtain immune T cells for ex vivo-activation. 5) Subjects' T cells are stored frozen until after chemoradiotherapy is completed. 6) Following chemoradiotherapy Subjects are infused with activated effector T cells followed by a 10-day course of low-dose interleukin 2 (IL-2). 7) Subjects then proceed with post therapy surveillance.
  Interventions: Biological: TVI-Brain-1; Procedure: Standard of Care; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Biological: TVI-Brain-1 — Attenuated autologous cancer cells and activated autologous blood-derived t cells
  Arms: Interventional TVI-Brain-1 Autologous Vaccine and activated autologous blood-derived t cells
Procedure: Standard of Care — Surgery for tumor removal or debulking to minimize tumor burden
Radiation: Radiotherapy — Conformal radiotherapy consists of fractionated focal irradiation at a dose of 2 Gy per fraction given once daily five days per week (Monday through Friday) over a period of six weeks.
Drug: Temozolomide — All Subjects receive 75 mg/m2 of temozolomide daily beginning on the first day of radiotherapy and continuing until the completion of radiotherapy. Standard of care Subjects will also receive adjuvant temozolomide .
  Other Names: Chemotherapy

SUMMARY:
This randomized study is designed to compare the combination of TVI-Brain-1 immunotherapy and standard therapy compared to standard therapy alone as a treatment for newly diagnosed MGMT unmethylated glioblastoma patients. The patients' own cancer cells collected after surgery are combined into a vaccine to produce an immune response that significantly increases the number of cancer neoantigen-specific effector T cell precursors in the patient's body. These cancer neoantigen-specific T cells are harvested from the blood, subsequently stimulated and expanded, and infused back into the patient.

DETAILED DESCRIPTION:
This randomized study is designed to compare the combination of TVI-Brain-1 immunotherapy and standard therapy compared to standard therapy alone as a treatment for newly diagnosed MGMT unmethylated glioblastoma patients. The general procedures include the collection and testing of cancer tissue samples after surgery and chemoradiation therapy (radiation and temozolomide). For the patients randomized into the investigational study treatment group, they will also receive two vaccinations created from their own cancer cells, undergo leukapheresis to collect immune T-cells from their blood, and transfer of those activated effector T-cells after chemoradiation therapy. All patients are followed with MRIs at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed MGMT unmethylated glioblastoma multiforme (no prior treatment)
* Sufficient cancer tissue obtained to allow for manufacture of autologous cancer cell vaccines
* The attenuated autologous cancer cell product generated has satisfied the product release criteria as determined by the sponsor quality control department
* Medical history, physical examination and laboratory testing performed within approximately 7 days before enrollment revealing kidney and liver organ function within normal limits
* not currently receiving glucocorticoids and have been off glucocorticoids for at least 24 hours prior to vaccination as well as when they receive the T cell infusion.
* Patient function assessment (Karnofsky score is > 60)
* a life expectancy of > 12 weeks.
* Hemoglobin is > 10 g/dL (may be transfused)
* White blood cell count is > 3,000 cells/microliter (mcL) of blood.
* Platelet count is > 100,000 platelets per mcL of blood (transfusion independent)
* Lymphocyte count is > 1,000 cells/mcL of blood.

Exclusion Criteria:

* another concomitant life-threatening disease (not including glioblastoma multiforme)
* a second malignancy that is not in remission as determined by the clinical investigator. Exception: squamous or basal cell carcinoma of the skin.
* requirement for treatment with glucocorticoids to control brain swelling
* presence of active autoimmune disease that is currently being actively treated.
* psychological, familial, sociological or geographical conditions that do not permit adequate medical follow-up and compliance with the study protocol.
* Current pregnancy or a plan to become pregnant within 1-year following the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Survival | From date of randomization until the date of death from any cause assessed up to 24 months after randomization.
  All Subjects will be evaluated and contacted to evaluate their status

SECONDARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression assessed up to 24 months after randomization
  Time to progression is evaluated by review and analysis of serial MRI's taken at specific Time to progression is evaluated by review and analysis of serial MRI's taken at specific timepoints

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 2 years
  Assessment of changes in patient through Physical Examination
Immunogenicity | Assessed at 24 hours after each vaccine administration
  Delayed-type hypersensitivity (DTH) skin testing using attenuated autologous cancer cells will be performed to assess the immunogenicity of the Subject's cancer.
Other genetic and immunologic parameters | Assessed at 24 hours after each vaccine administration
  The study is also designed to determine whether a wide variety of genetic and immunologic parameters that are monitored during and following treatment correlate with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jean Aguiar, APRN, Study Director — TVAX Biomedical, Inc
Locations (8):
- United States (8):
  - Center for Neurosciences, Tucson, Arizona
  - Cedar-Sanai Medical Center, Los Angeles, California
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Aaron Mammoser, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Capital Health, Pennington, New Jersey
  - Providence St. Vincent, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holladay FP, Heitz T, Chen YL, Chiga M, Wood GW. Successful treatment of a malignant rat glioma with cytotoxic T lymphocytes. Neurosurgery. 1992 Sep;31(3):528-33. doi: 10.1227/00006123-199209000-00015. PMID 1407433
- [Background] Holladay FP, Heitz T, Wood GW. Antitumor activity against established intracerebral gliomas exhibited by cytotoxic T lymphocytes, but not by lymphokine-activated killer cells. J Neurosurg. 1992 Nov;77(5):757-62. doi: 10.3171/jns.1992.77.5.0757. PMID 1403119
- [Background] Plautz GE, Touhalisky JE, Shu S. Treatment of murine gliomas by adoptive transfer of ex vivo activated tumor-draining lymph node cells. Cell Immunol. 1997 Jun 15;178(2):101-7. doi: 10.1006/cimm.1997.1140. PMID 9225000
- [Background] Sloan AE, Dansey R, Zamorano L, Barger G, Hamm C, Diaz F, Baynes R, Wood G. Adoptive immunotherapy in patients with recurrent malignant glioma: preliminary results of using autologous whole-tumor vaccine plus granulocyte-macrophage colony-stimulating factor and adoptive transfer of anti-CD3-activated lymphocytes. Neurosurg Focus. 2000 Dec 15;9(6):e9. doi: 10.3171/foc.2000.9.6.10. PMID 16817692
- [Background] Wood GW, Turner T, Wang YY, Holladay FP. Immune rejection of intracerebral gliomas using lymphocytes from glioma-bearing rats. J Immunother. 1999 Nov;22(6):497-505. doi: 10.1097/00002371-199911000-00004. PMID 10570748

DOCUMENTS (1):
  • Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT05685004/ICF_000.pdf